CLINICAL TRIAL: NCT00017095
Title: First Prospective Intergroup Translational Research Trial Assessing the Potential Predictive Value of p53 Using a Functional Assay in Yeast in Patients With Locally Advanced/Inflammatory or Large Operable Breast Cancer Prospectively Randomised to a Taxane Versus a Non Taxane Regimen
Brief Title: Biomarker (p53 Gene) Analysis and Combination Chemotherapy Followed by Radiation Therapy and Surgery in Treating Women With Large Operable or Locally Advanced or Inflammatory Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Swedish Breast Cancer Group (Other); Swiss Cancer Institute (Other); Anglo Celtic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-10994-p53; EORTC-10994; ACCOG-EORTC-10994; SAKK-EORTC-10994; SBGC-EORTC-10994; BIG-1-00
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; Microarray Analysis; Immunohistochemistry; Biopsy; Neoadjuvant Therapy; Radiotherapy

ARMS (2):
- non taxane based chemotherapy (Active Comparator): either FEC 100 or Canadian CEF or Tailored FEC for 6 cycles
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: epirubicin hydrochloride; Drug: fluorouracil; Genetic: microarray analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: biopsy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy
- taxane based chemotherapy (Experimental): Docetaxel for 3 cycles followed by Epirubicin/Docetaxel for 3 cycles
  Interventions: Drug: docetaxel; Drug: epirubicin hydrochloride; Genetic: microarray analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: biopsy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
  Arms: non taxane based chemotherapy
Drug: cyclophosphamide
  Arms: non taxane based chemotherapy
Drug: docetaxel
  Arms: taxane based chemotherapy
Drug: epirubicin hydrochloride
Drug: fluorouracil
  Arms: non taxane based chemotherapy
Genetic: microarray analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Currently patients with breast cancer are treated with one of several very similar combinations of drugs. Analysis of biomarkers in tumor tissue may help doctors predict how well patients with breast cancer will respond to treatment and help doctors choose the best drug regimen to treat each patient.

PURPOSE: This randomized phase III trial is studying giving different regimens of chemotherapy and comparing how well they work in treating women with large operable or locally advanced or inflammatory breast cancer. This study is also looking at whether analyzing a specific biomarker (p53) in tumor tissue may help doctors predict how well patients will respond to treatment and help doctors choose the best drug to treat each patient.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare neoadjuvant fluorouracil, epirubicin, and cyclophosphamide vs docetaxel and epirubicin followed by radiotherapy and surgery in women with locally advanced, inflammatory, or large operable breast cancer.
* Assess overall differences between the two arms.
* Assess interaction between p53 status and outcomes in each arm.
* Compare the progression-free survival of patients treated with these regimens.

Secondary

* Compare the distant metastasis-free survival and survival of patients treated with these regimens.
* Compare the clinical and pathological responses to these regimens in these patients.
* Compare the toxicity of these regimens in these patients.

Translational

* Determine the p53 status in order to study the treatment effect in each of the p53 subgroups and test the interaction between treatment and p53 status.
* Assess the level of agreement between p53 assessment by IHC method and functional test in yeast.
* Evaluate the prognostic and predictive value of "high risk" p53 mutations.
* Perform a survival analysis according to gene clusters defined with the use of microarrays.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to stage of disease (large T2-3 vs locally advanced or inflammatory), p53 status (negative vs positive vs unknown), and participating center. Patients are randomized to 1 of 2 chemotherapy treatment arms.

* Arm I (non-taxane arm): Patients receive 1 of 3 chemotherapy regimens comprising fluorouracil, epirubicin, and cyclophosphamide (FEC) (according to participating institution).

  * FEC 100: Patients receive fluorouracil IV over 15 minutes, epirubicin IV over 1 hour, and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Canadian FEC: Patients receive oral cyclophosphamide on days 1-14 and epirubicin IV and fluorouracil IV on days 1 and 8. If oral medications are not tolerated, patients may switch to cyclophosphamide IV on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Tailored FEC: Patients receive fluorouracil IV over 15 minutes, epirubicin IV over 1 hour, and cyclophosphamide IV over 1-2 hours on day 1. Patients also receive filgrastim (G-CSF) subcutaneously on days 2-15 or until blood counts recover. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (taxane arm): Patients receive docetaxel IV over 1 hour on days 1, 22, and 43 followed by epirubicin IV over 15 minutes and docetaxel IV over 1 hour on days 64, 85, and 106 in the absence of disease progression or unacceptable toxicity.

Following chemotherapy, patients may undergo loco-regional therapy comprising radiotherapy with or without breast conservation surgery or mastectomy. Patients with estrogen- and/or progesterone-receptor-positive disease also receive tamoxifen or an aromatase inhibitor for 5 years.

Two tumor samples (incisional or tricut biopsies) are taken before chemotherapy. Samples are analyzed by IHC, a functional test in yeast, and microarray analysis.

Patients are followed every 3 months for 1 year, every 4 months for 1.5 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 1,850 patients will be accrued for this study within 5.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Locally advanced or inflammatory disease

    * T4a-d, any N, M0 OR
    * Any T, N2 or N3, M0
    * Large operable T2 or T3 tumors
* No bilateral breast cancer
* Frozen tumor sample available

  * 1 incisional biopsy OR
  * 2 trucut biopsies from a 14G needle
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 70 and under

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.2 mg/dL
* SGOT less than 60 IU/L

Renal:

* Creatinine less than 1.35 mg/dL

Cardiovascular:

* LVEF normal by echocardiography or MUGA

Other:

* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No serious uncontrolled medical condition
* No uncontrolled psychiatric or addictive disorders
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1856 (Actual)
Dates: Start 2001-03; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | from randomization till first evidence of progression

SECONDARY OUTCOMES:
Distant metastasis-free survival | randomization till first evidence recurrence
Overall survival | randomization till death
Clinical and pathological responses | after 3rd and 6d cycle of chemotherapy
Clinical response according to RECIST criteria without pathologic response | after 3rd and 6d cycle of chemotherapy
Toxicity according to CTC v2.0 | from randomization
Agreement between p53 assessment by IHC method and functional test in yeast by analyzing the correlation between p52 and tumor status after 3 and 6 cycles of chemotherapy | after 3 and 6 cycles of chemotherapy
Tumor assessment using cDNA microarray technology | end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Herve Bonnefoi, Study Chair — Institut Bergonie, Bordeaux
Locations (39):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- France (10):
  - Centre Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Portugal (2):
  - Hospitais da Universidade de Coimbra (HUC), Coimbra
  - Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- Sweden (7):
  - Sahlgrenska University Hospital at Gothenburg University, Gothenburg (Goteborg)
  - Lund University Hospital, Lund
  - Malmo University Hospital, Malmo
  - Sahlgrenska University Hospital - Molndal at Gothenburg University, Mölndal
  - Orebro University Hospital, Örebro
  - Karolinska University Hospital - Huddinge, Stockholm
  - Uppsala University Hospital, Uppsala
- Switzerland (6):
  - Kantonspital Aarau, Aarau
  - Swiss Institute for Applied Cancer Research, Bern
  - Inselspital Bern, Bern
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - UniversitaetsSpital Zuerich, Zurich
- United Kingdom (5):
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Royal South Hants Hospital, Southampton, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Scottish Cancer Therapy Network, Edinburgh, Scotland

REFERENCES:
- [Background] Bonnefoi H, Potti A, Delorenzi M, Mauriac L, Campone M, Tubiana-Hulin M, Petit T, Rouanet P, Jassem J, Blot E, Becette V, Farmer P, Andre S, Acharya CR, Mukherjee S, Cameron D, Bergh J, Nevins JR, Iggo RD. Retraction--Validation of gene signatures that predict the response of breast cancer to neoadjuvant chemotherapy: a substudy of the EORTC 10994/BIG 00-01 clinical trial. Lancet Oncol. 2011 Feb;12(2):116. doi: 10.1016/S1470-2045(11)70011-0. No abstract available. PMID 21277543
- [Background] Desmedt C, Di Leo A, de Azambuja E, Larsimont D, Haibe-Kains B, Selleslags J, Delaloge S, Duhem C, Kains JP, Carly B, Maerevoet M, Vindevoghel A, Rouas G, Lallemand F, Durbecq V, Cardoso F, Salgado R, Rovere R, Bontempi G, Michiels S, Buyse M, Nogaret JM, Qi Y, Symmans F, Pusztai L, D'Hondt V, Piccart-Gebhart M, Sotiriou C. Multifactorial approach to predicting resistance to anthracyclines. J Clin Oncol. 2011 Apr 20;29(12):1578-86. doi: 10.1200/JCO.2010.31.2231. Epub 2011 Mar 21. PMID 21422418
- [Result] Bonnefoi H, Piccart M, Bogaerts J, Mauriac L, Fumoleau P, Brain E, Petit T, Rouanet P, Jassem J, Blot E, Zaman K, Cufer T, Lortholary A, Lidbrink E, Andre S, Litiere S, Lago LD, Becette V, Cameron DA, Bergh J, Iggo R; EORTC 10994/BIG 1-00 Study Investigators. TP53 status for prediction of sensitivity to taxane versus non-taxane neoadjuvant chemotherapy in breast cancer (EORTC 10994/BIG 1-00): a randomised phase 3 trial. Lancet Oncol. 2011 Jun;12(6):527-39. doi: 10.1016/S1470-2045(11)70094-8. Epub 2011 May 11. PMID 21570352
- [Result] Bonnefoi HR, Bogaerts J, Piccart M, et al.: Phase III trial (EORTC 10994/BIG 00-01) assessing the value of p53 using a functional assay to predict sensitivity to a taxane versus nontaxane primary chemotherapy in breast cancer: final analysis. [Abstract] J Clin Oncol 28 (Suppl 18): A-LBA503, 2010.
- [Result] Collingridge D. Expression of concern--validation of gene signatures that predict the response of breast cancer to neoadjuvant chemotherapy: a substudy of the EORTC 10994/BIG 00-01 clinical trial. Lancet Oncol. 2010 Sep;11(9):813-4. doi: 10.1016/S1470-2045(10)70185-6. Epub 2010 Jul 26. No abstract available. PMID 20667781
- [Result] Bonnefoi H, Zimmer AS, Piccart M, et al.: P53 functional assay in yeast: evaluation in 1856 patients in a large prospective clinical trial: EORTC 10994/BIG 00-01. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-1067, 2008.
- [Result] Bonnefoi H, Potti A, Delorenzi M, Mauriac L, Campone M, Tubiana-Hulin M, Petit T, Rouanet P, Jassem J, Blot E, Becette V, Farmer P, Andre S, Acharya CR, Mukherjee S, Cameron D, Bergh J, Nevins JR, Iggo RD. Validation of gene signatures that predict the response of breast cancer to neoadjuvant chemotherapy: a substudy of the EORTC 10994/BIG 00-01 clinical trial. Lancet Oncol. 2007 Dec;8(12):1071-1078. doi: 10.1016/S1470-2045(07)70345-5. Epub 2007 Nov 19. PMID 18024211 (Retraction: PMID 21277543 Bonnefoi H, Potti A, Delorenzi M, Mauriac L, Campone M, Tubiana-Hulin M, Petit T, Rouanet P, Jassem J, Blot E, Becette V, Farmer P, André S, Acharya CR, Mukherjee S, Cameron D, Bergh J, Nevins JR, Iggo RD. Lancet Oncol. 2011 Feb;12(2):116)
- [Result] Karina M, Bogaerts J, Piccart M, et al.: Preliminary safety data of the EORTC 10994/BIG 00-01 neoadjuvant trial comparing 3 cycles of docetaxel followed by 3 cycles of epirubicin-docetaxel versus 6 cycles of FEC 100 in patients with locally advanced/inflammatory or large operable breast cancer. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-3067, S146-7, 2006.
- [Result] Bonnefoi H, Farmer P, Delorenzi M, et al.: Is there a regimen-specific gene signature predicting for pathological complete response after neoadjuvant chemotherapy in hormone-negative breast cancer patients? A microarray substudy of 101 patients included in EORTC 10994/BIG 00-01 trial. [Abstract] Breast Cancer Research and Treatment 94 (Suppl 1): A-1040, 2005.
- [Result] Farmer P, Iggo R, Becette V, et al.: High quality gene expression microarray data from a multicentre prospective trial: results of the first microarray analysis in the EORTC 10994/ BIG 00-01 study. [Abstract] Eur J Cancer 2 (Suppl 3): A-155, 99, 2004.
- [Derived] Chatzipli A, Bonnefoi H, MacGrogan G, Sentis J, Cameron D, Poncet C; EORTC 10994/BIG 1-00 Consortium; Iggo R. Patterns of genomic change in residual disease after neoadjuvant chemotherapy for estrogen receptor-positive and HER2-negative breast cancer. Br J Cancer. 2021 Nov;125(10):1356-1364. doi: 10.1038/s41416-021-01526-3. Epub 2021 Sep 3. PMID 34480095
- [Derived] Bonnefoi H, Litiere S, Piccart M, MacGrogan G, Fumoleau P, Brain E, Petit T, Rouanet P, Jassem J, Moldovan C, Bodmer A, Zaman K, Cufer T, Campone M, Luporsi E, Malmstrom P, Werutsky G, Bogaerts J, Bergh J, Cameron DA; EORTC 10994/BIG 1-00 Study investigators. Pathological complete response after neoadjuvant chemotherapy is an independent predictive factor irrespective of simplified breast cancer intrinsic subtypes: a landmark and two-step approach analyses from the EORTC 10994/BIG 1-00 phase III trial. Ann Oncol. 2014 Jun;25(6):1128-36. doi: 10.1093/annonc/mdu118. Epub 2014 Mar 11. PMID 24618153